CLINICAL TRIAL: NCT03216213
Title: Evaluating Attitudes Towards Organ Donation in Singapore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HSS-1502-P02
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Control; Behavior
MeSH Terms: conditions — Behavior | interventions — Reading Frames

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Vignette contains no extra information
- Frame (Experimental): Vignette is framed in a particular manner
  Interventions: Other: Frame
- Norms (Experimental): Vignette contains extra information about norms
  Interventions: Other: Norms
- All (Experimental): Vignette contains extra information about norms and is framed in a particular manner.
  Interventions: Other: Frame; Other: Norms

INTERVENTIONS:
Other: Frame — Vignette is framed in a way that nudges participant to leave a legacy
  Arms: All; Frame
Other: Norms — Vignette informs the participant that most people choose an option to try to nudge participant into choosing that option as well
  Arms: All; Norms

SUMMARY:
One survey is conducted. Exploring the effect of different messages on family members' decision making on organ donation.

DETAILED DESCRIPTION:
The investigators intend to examine the impact of nudging interventions in the form of a vignette designed to emulate the standard procedure of informing family members of a loved one's unfavourable prognosis. The investigators intend to examine the effect of the interventions on the eventual decision-making process of the family member.

ELIGIBILITY:
Inclusion Criteria:

* Above age 21
* Singapore Citizens and Permanent Residents

Exclusion Criteria:

* Below age 21
* Non-citizens
* Not able to make decisions for self

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Binary survey item - Preferred option for mother's situation | 3 minutes
  A binary choice between 'Turning off life support' and 'Wait and see' which measures the efficacy of nudges on ultimate decision-making.
10cm line scale survey item - Willingness for participant's mother's organs to be donated under brain death | 3 minutes
  A 10cm line scale will be given and participants will be asked to put a cross on the line that corresponds to what they are feeling. This will measure their willingness for their mother's organs to be donated under the conditions of brain death.

SECONDARY OUTCOMES:
10cm line scale survey item - Willingness for participant's mother's organs to be donated under cardiac death | 3 minutes
  A 10cm line scale will be given and participants will be asked to put a cross on the line that corresponds to what they are feeling. This will measure their willingness for their mother's organs to be donated under the conditions of cardiac death.
10cm line scale survey item - Willingness for participant's own organs to be donated under brain death | 3 minutes
  A 10cm line scale will be given and participants will be asked to put a cross on the line that corresponds to what they are feeling. This will measure their willingness to donate their own organs under conditions of brain death.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided